CLINICAL TRIAL: NCT02513186
Title: A Dose Escalation, Safety, Pharmacokinetic, Pharmacodynamic and Preliminary Efficacy Study of SAR650984 (Isatuximab) Administered Intravenously in Combination With Bortezomib - Based Regimens in Adult Patients With Newly Diagnosed Multiple Myeloma Non Eligible for Transplantation or No Intent for Immediate Transplantation
Brief Title: Study of Isatuximab Combined With Bortezomib + Cyclophosphamide + Dexamethasone (VCD) and Bortezomib + Lenalidomide + Dexamethasone (VRD) in Newly Diagnosed Multiple Myeloma (MM) Non Eligible for Transplant or No Intent for Immediate Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD13983; U1111-1154-6102 (Registry Identifier: ICTRP); 2014-001251-23 (EudraCT Number)
Record Dates: First submitted 2015-07-16; First posted 2015-07-31 (Estimated); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Plasma Cell Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib; Cyclophosphamide; Dexamethasone; isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isatuximab (Experimental): VCDI cohort: Isatuximab (escalating dose) + bortezomib + cyclophosphamide + dexamethasone (VCDI): Induction phase will be 50 weeks (12 cycles). The duration of a cycle will be 42 days (6 weeks) for Cycle 1 (C1) and 28 days (4 weeks) for subsequent cycles. The duration of a cycle of the maintenance phase will be 28 days (4 weeks). After C12, isatuximab will be administered at its initial assigned dose and dexamethasone once every 28 days.
  VRDI cohort parts A and B: Isatuximab + bortezomib + dexamethasone + lenalidomide (VRDI): Induction phase will be 24 weeks (4 cycles at 6 weeks/cycle). The duration of a cycle of the maintenance phase will be 28 days (4 weeks). Maintenance therapy may continue until disease progression, unacceptable AE or patient willingness to discontinue.
  VRDI Part A: Enrollment to begin after the VCDI cohort is completed.
  VRDI Part B: Enrollment to begin after the VRDI part A is completed.
  Interventions: Drug: lenalidomide; Drug: bortezomib; Drug: cyclophosphamide; Drug: dexamethasone; Drug: isatuximab SAR650984

INTERVENTIONS:
Drug: lenalidomide — Pharmaceutical form: tablet Route of administration: oral
  Other Names: Revlimid
Drug: bortezomib — Pharmaceutical form: lyophilized powder for subcutaneous injection Route of administration: subcutaneous
  Other Names: Velcade
Drug: cyclophosphamide — Pharmaceutical form: tablet Route of administration: oral
  Other Names: Endoxan
Drug: dexamethasone — Pharmaceutical form: tablet or solution for infusion Route of administration: oral or intravenous
Drug: isatuximab SAR650984 — Pharmaceutical form: solution for infusion Route of administration: intravenous
  Other Names: Sarclisa

SUMMARY:
Primary Objectives:

* VCDI cohort:

  * To determine the maximum tolerated dose (MTD) and recommended dose (RD) of SAR650984 isatuximab when administered in combination with bortezomib (Velcade®) , cyclophosphamide, and dexamethasone (VCDI) based on the dose-limiting toxicity(ies) (DLTs) observed in patients with newly diagnosed multiple myeloma non-eligible for transplantation
  * To evaluate safety and preliminary efficacy (overall response rate and complete response rate) of isatuximab administered at the selected dose in combination with bortezomib based regimin VCDI according to IMWG criteria.
* VRDI Part A cohort and Part B cohort:

  * To evaluate the preliminary efficacy (complete response [CR] rate) of isatuximab administered at the selected dose in combination with bortezomib based regimen: VRDI, (bortezomib, lenalidomide, dexamethasone) according to IMWG criteria in adult patients with newly diagnosed MM non eligible for transplantation or no intent for immediate transplantation.

Secondary Objectives:

* VCDI cohort:

  * To characterize the overall safety profile of SAR650984 in combination with VCD regimen, including cumulative toxicities.
  * To characterize the pharmacokinetic (PK) profile of SAR650984/isatuximab and each combination drug in VCDI regimen.
  * To evaluate the immunogenicity of SAR650984 in combination treatments.
  * To evaluate the preliminary efficacy of VCDI regimen in terms of duration of response and progression-free survival.
  * To assess the relationship between clinical effects (adverse event [AE] and/or tumor response) and CD38 receptor density.
* VRDI Part A cohort and Part B cohort:

  * To characterize the overall safety profile of isatuximab in combination with VRD regimen.
  * To evaluate the infusion duration (only applicable for VRDI Part B cohort)
  * To characterize the PK profile of isatuximab and each combination drug in VRDI regimen.
  * To evaluate the immunogenicity of isatuximab in combination treatments.
  * To evaluate the preliminary efficacy of VRDI regimen in terms of ORR, DOR, and PFS.
  * To evaluate the impact of M protein measurement without isatuximab interference (via the SEBIA HYDRASHIFT 2/4 isatuximab IFE test) on CR and BOR assessment.
  * To assess the relationship between clinical effects (AE and/or tumor response) and CD38 receptor density (only applicable for VRDI Part A cohort).
  * To assess MRD negativity rate in patients achieving a CR or VGPR and explore correlation with clinical outcome.

DETAILED DESCRIPTION:
The duration of the study for an individual patient will include:

* A period to assess eligibility (screening or baseline period) of up to 3 weeks for VCDI cohort, up to 28 days for VRDI cohort;
* for patients in the VCDI cohort: a treatment period including up to 12 induction treatment cycles (50-week duration).
* for patients in the VRDI cohort: a treatment period including up to 4 induction cycles (24 week duration).
* Following induction, both cohorts have maintenance periods consisting of 4 week cycles until progression, unacceptable AE, or patient willingness to discontinue and an end-of-treatment visit at least 30 days following the last administration of treatment.
* Patients that discontinue therapy for reasons other than progression will have follow-up visits until progression or until the patient receives another anticancer therapy, whichever is earlier.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed patients with measurable multiple myeloma defined as at least one of the following:

  * Serum M protein ≥1 g/dL (≥10 g/L).
  * Urine M protein ≥200 mg/24 hours.
  * Serum free light chain (sFLC) assay: involved free light chain assay ≥10 mg/dL (≥100 mg/L) and an abnormal sFLC ratio (<0.26 or >1.65).
* Patients with ultra-high risk smoldering multiple myeloma fulfilling the International Myeloma Working Group criteria are eligible.
* Patient is not eligible for transplant.
* Patient with no intent for immediate transplant as per investigator's decision are also eligible for VRDI Part B cohort only.

Exclusion criteria:

* Eastern Cooperative Oncology Group performance status >2.
* Poor bone marrow reserve.
* Poor organ function.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Assessment of dose-limiting toxicities (DLTs) in VCDI cohort | Up to 6 weeks per treated patient
Overall response rate (VCDI) | Up to 34 weeks of treatment (induction phase)
Complete response rate (VCDI) | Up to 34 weeks of treatment (induction phase)
Complete response rate (VRDI) | Up to 104 weeks of treatment (induction and maintenance phase) in VRDI part A and part B cohorts

SECONDARY OUTCOMES:
Number of patients with adverse events (AEs), clinically significant changes in laboratory tests and vital signs according to the National Cancer Institute - Common Toxicity Criteria (NCI-CTC) version 4.03 grade scaling | VCDI: Up to approximately 106 weeks, VRDI Part A and Part B: Up to approximately 104 weeks
Overall response rate (VRDI) | Up to 104 weeks of treatment (induction and maintenance phase) in VRDI part A and part B cohorts
Infusion duration | VRDI Part B: Up to 104 weeks of treatment
Assessment of PK parameter: Partial area under the serum concentration time curve (AUC) | VCDI: Up to approximately 42 weeks, VRDI: Up to approximately 48 weeks
Assessment of PK parameter: Maximum observed concentration (Cmax) | VCDI: Up to approximately 42 weeks, VRDI: Up to approximately 48 weeks
Levels of human antidrug antibodies (ADA) | VCDI: Up to approximately 42 weeks, VRDI: Up to approximately 48 weeks
Duration of response - time | VCDI and VRDI: Until treatment discontinuation by the last patient
Progression-free survival for VCDI | VCDI: 30 months after LPI
Progression-free survival for VRDI | VRDI Part A and Part B: 24 months after LPI
MRD negativity rate | Up to 3 years of treatment (induction and maintenance phase) in VRDI part A and part B cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (12):
- France (3):
  - Investigational Site Number : 250002, Nantes
  - Investigational Site Number : 250003, Pierre-Bénite
  - Investigational Site Number : 250001, Toulouse
- Germany (2):
  - Investigational Site Number : 276003, Berlin
  - Investigational Site Number : 276002, Leipzig
- Italy (3):
  - Investigational Site Number : 380003, Milan
  - Investigational Site Number : 380002, Roma
  - Investigational Site Number : 380001, Torino
- Spain (4):
  - Investigational Site Number : 724004, Santander, Cantabria
  - Investigational Site Number : 724001, Pamplona, Navarre
  - Investigational Site Number : 724003, Madrid
  - Investigational Site Number : 724002, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Ocio EM, Perrot A, Bories P, San-Miguel JF, Blau IW, Karlin L, Martinez-Lopez J, Wang SY, Bringhen S, Marcatti M, Mateos MV, Rodriguez-Otero P, Oliva S, Nogai A, Le Roux N, Dong L, Mace S, Gassiot M, Fitzmaurice T, Oprea C, Moreau P. Efficacy and safety of isatuximab plus bortezomib, lenalidomide, and dexamethasone in patients with newly diagnosed multiple myeloma ineligible/with no immediate intent for autologous stem cell transplantation. Leukemia. 2023 Jul;37(7):1521-1529. doi: 10.1038/s41375-023-01936-7. Epub 2023 Jun 14. PMID 37316728